CLINICAL TRIAL: NCT04141202
Title: Structured Physical Exercise in Short-term Inpatient Treatment of Substance Use Disorder: Implications for Abstinence, Quality of Life, Physical- and Mental Health
Brief Title: Structured Physical Exercise in Short-term Inpatient Treatment of Substance Use Disorder
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/501
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Substance-Related Disorders; Drug Abuse; Drug Dependence
Keywords: Exercise therapy; Exercise physiology
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exercise group

SUMMARY:
In 2017, structured physical exercise with high intensity was implemented as a part of the treatment program at St. Olav Hospital Clinic of Substance Use and Addiction Medicine.

The objective of this study is to examine whether implementing structured physical exercise in the treatment program has implications for patients' physical and mental health and quality of life after completing a 3 month residential treatment program.

The results of this study will benefit substance use disorder patients in the future, and may have an impact on further implementation of physical exercise in addiction treatment clinics both nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Being an inpatient at the clinic

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with substance use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Physical health | 18 months
  Change in oxygen uptake
Physical health | 18 months
  Change in maximum leg strength
Mental health | 18 months
  assessed by a in-house developed questionnaire, which is composed of 4 parts: Severity of Dependence 5-items (each of the five items is scored on a 4-point scale (0-3). Total score is the sum of the 5-item ratings. The higher the score the higher the level of dependence); Circumstances, Motivation, Readiness, and Suitability instrument (Five items measured on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (totally agree). High scores indicate increased intrinsic motivation); Quality-of-Life rating five items recorded on a five-point Likert scale: 1 (very poor) - 5 (very good). The raw scores are transformed to a decimal scale, ranging from 0.1 worst score to 0.9 best score); Hopkins Symptom Checklist (HSCL-10): Ten items recorded on a four-point Likert scale: (1) not at all - (4) extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Smedsrud, Study Director — St Olavs Hospital Klinikk for rus- og avhengighetsmedisin
Locations (1):
- St Olavs Hospital HF Klinikk for rus og avhengighetsmedisin, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No